CLINICAL TRIAL: NCT03667534
Title: Dry Blood Spot Screening Test for Neonatal Cholestasis Patients
Acronym: DBS-SCReNC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201804007RIND
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Cholestasis in Newborn Infant; Biliary Atresia
Keywords: cholestasis; new born screening; dry blood spot; biliary atresia
MeSH Terms: conditions — Biliary Atresia; Cholestasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood serum sample and urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dry blood spot screening — Dry blood spot measurement of biomarker for screening of cholestasis patients

SUMMARY:
Cholestatic jaundice with multitude of causes affects approximately 1 in every 2,500 infants. Of the many conditions that cause neonatal cholestasis, the most commonly identifiable are biliary atresia (BA) (25%-35%). The incidence in Taiwan was 1.2 to 2.0 per 10,000 live birth. Prognosis and survival are improved if bile drainage is restored by a Kasai portoenterostomy. Stool color card was introduced to Taiwan in 2002 and national screening program was started in 2004. The rate of age at Kasai operation <60 days improved from 49.4% before year 2002 to 65.7% after introducing nationwide stool color card screening in Taiwan. There was a great improvement in early diagnosis for biliary atresia after stool color card screening and there were still many researches tried to improve the timing of diagnosis. A prospective cohort observational study on neonates under 27 days old at London showed that serum conjugated bilirubin > 18 micromol/l in plasma measured at 6-10 days is a reliable marker for neonatal cholestasis liver disease with sensitivity 100%, specificity 99.59% (95% CI 99.5-99.67), PPV 10.3% (95% CI 4.50-16.0).

Our study aims to developed a screening test for neonatal cholestasis using dry blood spot to improve patient survival by early diagnosis of treatable neonatal cholestasis disease, such as biliary atresia and inborn error of bile acid metabolism. The diseases markers for neonatal cholestasis we aims including basic clinical blood test examination profiles, inflammatory markers, fibrosis markers, immune profiles. In phase I study we will enroll cholestasis patients at National Taiwan University Children Hospital. We will collect patients' blood on dry blood spot and measure the disease markers for cholestasis disease. In phase II study, we will enroll the cholestasis patients and healthy newborn without cholestasis. We will review their newborn screening at 3 days old. Newborn screening dry blood spot will be examined for the disease markers and compared with healthy control without cholestasis. ROC curve analysis will be performed to find the best cut-off to screen for neonatal cholestasis patients.

The findings will aid early diagnosis in the patients and hence improve the survival.

DETAILED DESCRIPTION:
Aims:

1. Developed a screening test for neonatal cholestasis using dry blood spot
2. Improve patient survival by early diagnosis of treatable neonatal cholestasis disease such as biliary atresia and inborn error of bile acid metabolism.

Phase I - Validation of method for quantification of disease markers on dry blood spot.

Pediatric children with cholestasis diagnose at National Taiwan University Hospital during admission or out-patient clinic will be collected for the Phase I study. 5ml of venous blood will be collected for measurement of disease markers during routine follow-up at National Taiwan University Hospital outpatient clinic. Dried blood spot (DBS) specimens are collected from patients by applying a whole blood, drawn by lancet from the finger, heel or toe, a provided filter paper. To evaluate the stability of disease markers on DBS, a total 10 blood spots (each blood spout contain 50 - 75 microL of blood) will be applied on the filter paper at day 0. The collected blood spots samples of a single patient at day 0 will be evaluated at the day of DBS collection and followed by day 3, day 7, 6 months and 1 year after sample collection. The purpose of repeat measurement of single patient sample at different time point is to evaluate the possible effect of time effect on the accuracy of the data. 5 blood spots are separated and protected from light with a light blocking envelope to compare the light effect on disease markers degradation (Table 1). Serum disease markers measured with conventional method will be served as reference and compared with DBS samples at different time points. 30 patients will be collected to validate the correlation between serum and DBS disease markers level.

Phase II - Pilot study In the pilot study, we aim to develop dry blood spot method for the screening of neonatal cholestasis. Children with neonatal cholestasis disease previously diagnosed at Department of Pediatrics, National Taiwan University Children's Hospital from 2007 or newly diagnosed children will be recruited retrospectively from chart review. Patients with indirect type hyperbilirubinemia and healthy neonates will be enrolled as control. We will analyze neonatal cholestasis and control patients dry blood spot screening test after birth to quantify disease markers level. ROC curve analysis will be conducted on bilirubin quantity to find the best cutoff to screen for neonatal cholestasis. The sample size of case and control study is 20 cases and 20 controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with jaundice
* Healthy volunteers

Exclusion Criteria:

* Subjects who do not agree with study protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with jaundice and healthy volunteers are included for testing the efficacy and accuracy of the screening test.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-09-09 (Actual); Primary Completion 2021-06-08 (Estimated); Study Completion 2021-09-09 (Estimated)

PRIMARY OUTCOMES:
Cholestasis | on the time of enrollment
  Direct bilirubin > 1.0mg/dl or Direct bilirubin to total bilirubin ratio > 0.2

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwei Chang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No sharing plan